CLINICAL TRIAL: NCT04618562
Title: Impact of Revival Active Program on Adolescents With Depression: A Pilot Study
Brief Title: Revival Active Program for Adolescents With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revival Active (Other)
Collaborators: L.E.A.D (Unknown); NMP Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RAP/002
Record Dates: First submitted 2020-10-28; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Depression
Keywords: Adolescent; Revival Active Program
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Revival Active Program (Experimental): Revival Program included supervised play group, twice a week followed by home practice.
  Interventions: Other: Revival Active Program

INTERVENTIONS:
Other: Revival Active Program — Program comprised of physical activities, group play, mind games, reasoning and discussion on sleeted topics, breath work and relaxation techniques, 60 minutes all together.

SUMMARY:
Active play and sports has shown to be effective intervention in managing depression. Extending the support with Mind body therapy, Revival Active Program was designed as an early intervention for adolescents.

To measure the efficacy and feasibility of the community based revival active play intervention for adolescent depression, present pilot study was undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with depression as per the DSM IV-TR criteria
* Parents willing to give written informed consent

Exclusion Criteria:

* Physical limitation for active sports
* Co-morbid mental health diagnosis
* high risk of self harm/ suicide
* history of self harm or harming someone else

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Depression | Changes from baseline depression at 8-week
  Children Depression Inventory-II was used to assess depression level

SECONDARY OUTCOMES:
Self-Efficacy for Children | Changes from baseline self -efficacy at 8-week
  Emotional, social and academic self efficacy was assessed using Self-Efficacy Questionnaire for Children

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Patel, Study Director — Revival Active Limited; Tejal Patel, Study Director — Revival Active Limited; Sadhana Sharma, Study Chair — L.E.A.D; Sahil Signal, Principal Investigator — NMP Medical Research Institute, India
Locations (1):
- Gyansanjeevani, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided